CLINICAL TRIAL: NCT00158418
Title: Cemented Versus Uncemented Fixation of Humeral Components in Total Shoulder Arthroplasty for Osteoarthritis of the Shoulder
Brief Title: Cemented vs. Non-Cemented TSA for OA of the Shoulder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fowler Kennedy Sport Medicine Clinic (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Robert Litchfield, FKSMC
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FKSMC-CIHR-2; UCT-137451
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2009-01-29 (Estimated); Status verified 2005-09

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis; shoulder; randomized trial; cement
MeSH Terms: conditions — Osteoarthritis

INTERVENTIONS:
Procedure: Cemented Humeral Stem
Procedure: Uncemented Humeral Stem

SUMMARY:
The purpose of the study is to investigate the fixation of the humeral component in total shoulder arthroplasty for primary osteoarthritis of the glenohumeral joint.Our hypothesis is that uncemented fixation of the humerus will result in better disease-specific quality of life, decreased incidence of radiographic loosening, decrease operative time and no increase in complications.

DETAILED DESCRIPTION:
Currently, cement fixation of the humeral component is recommended as the standard of care and review of the literature indicates that this fixation is associated with a low complication rate. Uncemented fixation is promising in its potential to provide long-term, stable fixation yet comparative results to cemented stems are not available at this time.

Despite an absence of data to support their use, there has been an exponential increase in the use of uncemented humeral component fixation in shoulder arthroplasty. This push may be dictated by the desire to reduce operative time in an attempt to cut surgical expenses. This goal is particularly highlighted by the efforts of government and third party bodies to maximize return on limited funds. There is no conclusive clinical data at this time to suggest that uncemented fixation yields results that are better than cemented fixation in the shoulder.

This multi-centre, prospective, randomized double blinded clinical trial will compare cemented versus uncemented/tissue-ingrowth fixation of the humeral component in total shoulder arthroplasty. Patients are recruited from 10 centres across Canada by surgeons with extensive experience in total shoulder arthroplasty. Patients will be randomized to receive either a cemented or uncemented humeral stem. All other variables will be controlled for.

The main evaluation of patient outcome is disease-specific quality of life. Validated tools evaluating shoulder function are being used for this purpose, as required by various societies. These include the Western Ontario Osteoarthritis of the Shoulder Index (WOOS), the most responsive; Constant, preferred by European investigators; American Shoulder and Elbow Surgeons (ASES) Standardized Shoulder Assessment and Shoulder Score Index, preferred by the ASES. Overall global health status is measured using the SF-36. Several secondary outcomes are monitored for during the post-operative course. These are: shoulder function, radiographic evaluation of component fixation, operative time and the incidence of revision surgery and complications.

ELIGIBILITY:
Inclusion Criteria:

1. Primary osteoarthritis of the shoulder of grade III or higher (Kellgren and Lawrence modified for the shoulder
2. Patients who have failed standard conservative management of their shoulder osteoarthritis

Exclusion Criteria:

1. Patients with secondary OA resulting from major joint trauma, infection, avascular necrosis, cuff tear arthropathy, chronic dislocation, massive rotator cuff tear, inflammatory arthropathy, Charcot's arthropathy or previous shoulder surgery (other than arthroscopic debridement)
2. Patients with preoperative CT scans of the shoulder which show insufficient glenoid bone stock that would not allow for implantation of a glenoid prosthesis
3. Active joint or systemic infection
4. Significant muscle paralysis
5. Major medical illness (life expectancy less then 2yrs or unacceptably high operative risk)
6. Unable to speak or read English/French
7. Psychiatric illness that precludes informed consent
8. Unwilling to be followed for 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2002-08; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
disease specific quality of life comparing the 2 groups at 2 years using several shoulder function rating scales.
the Western Ontario Osteoarthritis of the Shoulder Index (WOOS)
the Constant Score
American Shoulder and Elbow Surgeons (ASES) Standardized Shoulder Assessment form.
Short Form-12

SECONDARY OUTCOMES:
the evaluation of radiolucent lines indicative of implant loosening
the incidence of revision surgery complications

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Litchfield, MD, FRCSC, Principal Investigator — Fowler Kennedy Sport Medicine Clinic
Locations (1):
- Fowler Kennedy Sport Medicine Clinic, London, Ontario, Canada

REFERENCES:
- [Background] Barrack RL, Castro F, Guinn S. Cost of implanting a cemented versus cementless femoral stem. J Arthroplasty. 1996 Jun;11(4):373-6. doi: 10.1016/s0883-5403(96)80025-8. PMID 8792242
- [Background] Brems JJ. Rehabilitation following total shoulder arthroplasty. Clin Orthop Relat Res. 1994 Oct;(307):70-85. PMID 7924050
- [Background] Brenner BC, Ferlic DC, Clayton ML, Dennis DA. Survivorship of unconstrained total shoulder arthroplasty. J Bone Joint Surg Am. 1989 Oct;71(9):1289-96. PMID 2793880
- [Background] Brown DD, Friedman RJ. Postoperative rehabilitation following total shoulder arthroplasty. Orthop Clin North Am. 1998 Jul;29(3):535-47. doi: 10.1016/s0030-5898(05)70027-4. PMID 9706298
- [Background] Cameron B, Galatz L, Williams GR Jr. Factors affecting the outcome of total shoulder arthroplasty. Am J Orthop (Belle Mead NJ). 2001 Aug;30(8):613-23. PMID 11520017
- [Background] Cofield RH, Daly PJ. Total shoulder arthroplasty with a tissue-ingrowth glenoid component. J Shoulder Elbow Surg. 1992 Mar;1(2):77-85. doi: 10.1016/S1058-2746(09)80124-9. Epub 2009 Feb 19. PMID 22959043
- [Background] Cofield RH. Total shoulder arthroplasty with the Neer prosthesis. J Bone Joint Surg Am. 1984 Jul;66(6):899-906. doi: 10.2106/00004623-198466060-00010. PMID 6736090
- [Background] Cofield RH. Uncemented total shoulder arthroplasty. A review. Clin Orthop Relat Res. 1994 Oct;(307):86-93. PMID 7924051
- [Background] Constant CR, Murley AH. A clinical method of functional assessment of the shoulder. Clin Orthop Relat Res. 1987 Jan;(214):160-4. PMID 3791738
- [Background] Cuomo F, Checroun A. Avoiding pitfalls and complications in total shoulder arthroplasty. Orthop Clin North Am. 1998 Jul;29(3):507-18. doi: 10.1016/s0030-5898(05)70025-0. PMID 9706296
- [Background] Fenlin JM Jr, Frieman BG. Indications, technique, and results of total shoulder arthroplasty in osteoarthritis. Orthop Clin North Am. 1998 Jul;29(3):423-34. doi: 10.1016/s0030-5898(05)70018-3. PMID 9706289
- [Background] Gartsman GM, Russell JA, Gaenslen E. Modular shoulder arthroplasty. J Shoulder Elbow Surg. 1997 Jul-Aug;6(4):333-9. doi: 10.1016/s1058-2746(97)90000-8. PMID 9285872
- [Background] Havig MT, Kumar A, Carpenter W, Seiler JG 3rd. Assessment of radiolucent lines about the glenoid. An in vitro radiographic study. J Bone Joint Surg Am. 1997 Mar;79(3):428-32. PMID 9070534
- [Background] Hawkins RJ, Bell RH, Jallay B. Total shoulder arthroplasty. Clin Orthop Relat Res. 1989 May;(242):188-94. PMID 2706849
- [Background] KELLGREN JH, LAWRENCE JS. Radiological assessment of osteo-arthrosis. Ann Rheum Dis. 1957 Dec;16(4):494-502. doi: 10.1136/ard.16.4.494. No abstract available. PMID 13498604
- [Background] Kelly JD Jr, Norris TR. Decision making in glenohumeral arthroplasty. J Arthroplasty. 2003 Jan;18(1):75-82. doi: 10.1054/arth.2003.50005. PMID 12555187
- [Background] Lo IK, Griffin S, Kirkley A. The development of a disease-specific quality of life measurement tool for osteoarthritis of the shoulder: The Western Ontario Osteoarthritis of the Shoulder (WOOS) index. Osteoarthritis Cartilage. 2001 Nov;9(8):771-8. doi: 10.1053/joca.2001.0474. PMID 11795997
- [Background] Laupacis A, Bourne R, Rorabeck C, Feeny D, Tugwell P, Wong C. Comparison of total hip arthroplasty performed with and without cement : a randomized trial. J Bone Joint Surg Am. 2002 Oct;84(10):1823-8. doi: 10.2106/00004623-200210000-00013. PMID 12377914
- [Background] Matsen FA 3rd. Early effectiveness of shoulder arthroplasty for patients who have primary glenohumeral degenerative joint disease. J Bone Joint Surg Am. 1996 Feb;78(2):260-4. doi: 10.2106/00004623-199602000-00013. PMID 8609117
- [Background] Matsen FA 3rd, Iannotti JP, Rockwood CA Jr. Humeral fixation by press-fitting of a tapered metaphyseal stem: a prospective radiographic study. J Bone Joint Surg Am. 2003 Feb;85(2):304-8. doi: 10.2106/00004623-200302000-00018. PMID 12571309
- [Background] McElwain JP, English E. The early results of porous-coated total shoulder arthroplasty. Clin Orthop Relat Res. 1987 May;(218):217-24. PMID 3568483
- [Background] Neer CS 2nd. Replacement arthroplasty for glenohumeral osteoarthritis. J Bone Joint Surg Am. 1974 Jan;56(1):1-13. No abstract available. PMID 4812164
- [Background] Neer CS 2nd, Watson KC, Stanton FJ. Recent experience in total shoulder replacement. J Bone Joint Surg Am. 1982 Mar;64(3):319-37. No abstract available. PMID 7061549
- [Background] Norris BL, Lachiewicz PF. Modern cement technique and the survivorship of total shoulder arthroplasty. Clin Orthop Relat Res. 1996 Jul;(328):76-85. doi: 10.1097/00003086-199607000-00014. PMID 8653982
- [Background] Richards RR, An KN, Bigliani LU, Friedman RJ, Gartsman GM, Gristina AG, Iannotti JP, Mow VC, Sidles JA, Zuckerman JD. A standardized method for the assessment of shoulder function. J Shoulder Elbow Surg. 1994 Nov;3(6):347-52. doi: 10.1016/S1058-2746(09)80019-0. Epub 2009 Feb 13. PMID 22958838
- [Background] Skirving AP. Total shoulder arthroplasty -- current problems and possible solutions. J Orthop Sci. 1999;4(1):42-53. doi: 10.1007/s007760050073. PMID 9914429
- [Background] Smith KL, Matsen FA 3rd. Total shoulder arthroplasty versus hemiarthroplasty. Current trends. Orthop Clin North Am. 1998 Jul;29(3):491-506. doi: 10.1016/s0030-5898(05)70024-9. PMID 9706295
- [Background] Torchia ME, Cofield RH, Settergren CR. Total shoulder arthroplasty with the Neer prosthesis: long-term results. J Shoulder Elbow Surg. 1997 Nov-Dec;6(6):495-505. doi: 10.1016/s1058-2746(97)90081-1. PMID 9437598
- [Background] Weinberger M, Tierney WM, Cowper PA, Katz BP, Booher PA. Cost-effectiveness of increased telephone contact for patients with osteoarthritis. A randomized, controlled trial. Arthritis Rheum. 1993 Feb;36(2):243-6. doi: 10.1002/art.1780360216. PMID 7679273
- [Background] Wirth MA, Rockwood CA Jr. Complications of shoulder arthroplasty. Clin Orthop Relat Res. 1994 Oct;(307):47-69. PMID 7924048
- [Background] Wirth MA, Agrawal CM, Mabrey JD, Dean DD, Blanchard CR, Miller MA, Rockwood CA Jr. Isolation and characterization of polyethylene wear debris associated with osteolysis following total shoulder arthroplasty. J Bone Joint Surg Am. 1999 Jan;81(1):29-37. doi: 10.2106/00004623-199901000-00005. PMID 9973051
- [Background] Kempf JF, Walch G, Lacaze F. Results of Shoulder Arthroplasty in Primary Glenohumeral Osteoarthritis. In Shoulder Arthroplasty. Springer-Verlag, Berlin, Germany, 1999, 203-210.
- [Background] Kirkley A, Litchfield R, Patterson S, Lo I. Hemi vs. Total Shoulder Arthroplasty in Primary Shoulder Osteoarthritis. Annual meeting of the Canadian Orthopaedic Association, Edmonton, Alberta, June 2000.
- [Background] Kreidie A.,Arthritis: a crisis for Canadians. Medical Post, May 16, 2000, pp 16.
- [Derived] Litchfield RB, McKee MD, Balyk R, Mandel S, Holtby R, Hollinshead R, Drosdowech D, Wambolt SE, Griffin SH, McCormack R. Cemented versus uncemented fixation of humeral components in total shoulder arthroplasty for osteoarthritis of the shoulder: a prospective, randomized, double-blind clinical trial-A JOINTs Canada Project. J Shoulder Elbow Surg. 2011 Jun;20(4):529-36. doi: 10.1016/j.jse.2011.01.041. PMID 21570660